CLINICAL TRIAL: NCT02574260
Title: Phase 2 Extension Protocol for Extended Use of OncoVEX^GM-CSF for Eligible Patients Participating in Study 002/03: Study of the Efficacy, Safety and Immunogenicity of OncoVEX^GM-CSF in Patients With Stage IIIc and Stage IV Malignant Melanoma
Brief Title: An Extension Protocol for the Extended Use of Talimogene Laherparepvec for Eligible Patients Who Participated in Study 002/03 (NCT00289016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioVex Limited (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002/03-E
Record Dates: First submitted 2015-09-18; First posted 2015-10-12 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Talimogene Laherparepvec (Experimental): Participants received talimogene laherparepvec 10⁸ plaque forming units (PFU)/mL (up to 4 mL depending on tumor size) administered intratumorally every 2 weeks, on Day 1 and Day 15 of 28-day cycles until discontinuation criteria were met.
  Interventions: Biological: Talimogene Laherparepvec

INTERVENTIONS:
Biological: Talimogene Laherparepvec — Administered by intratumoral injection.
  Other Names: OncoVEX^GM-CSF; T-VEC; IMLYGIC

SUMMARY:
The primary objective of this extension study was to further assess the safety and tolerability of talimogene laherparepvec. Secondary objectives were to assess objective tumor response rate and survival.

DETAILED DESCRIPTION:
This was an extension study to the multicenter, open-label, phase 2 Study 002/03 (NCT00289016). Participants who had received the maximum 24 treatments under Study 002/03 and met the inclusion and exclusion criteria were eligible to enroll.

Participants continued to receive talimogene laherparepvec until discontinuation criteria were met. The discontinuation criteria were complete response, clinically significant progressive disease that rendered further dosing futile, receipt of 24 treatments or 12 months on treatment (whichever was longer), occurrence of an unacceptable toxicity, death, investigator determination that other treatment was warranted, or another criterion for withdrawal from treatment (participant request, noncompliance with study procedures, or sponsor request).

ELIGIBILITY:
Inclusion Criteria:

1. Previously participated in Study 002/03 and met 1 of the following:

   1. Received the maximum 24 treatment injections in Study 002/03 and had not yet achieved a complete response (CR) and whose response to OncoVEX^GM-CSF indicated that treatment beyond 12 months was warranted, or
   2. Did achieve a CR in Study 002/03 and developed disease progression within 12 months of achieving a CR, or
   3. Terminated treatment in Study 002/03 to allow for treatment of brain metastases. Treatment for brain metastases was no longer ongoing and the patient was able to return to OncoVEX^GM-CSF injections within 3 months of completing treatment for brain metastases.
2. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.

Exclusion Criteria:

1. Prior Common Toxicity Criteria for Adverse Events (CTCAE) Grade 3 or 4 toxicity related to OncoVEX^GM-CSF of any organ system (with the exception of injection site reactions, fever and vomiting);
2. History of Grade 3 fatigue lasting > 1 week while on OncoVEX^GM-CSF treatment;
3. History of Grade 3 arthralgia/myalgias while on OncoVEX^GM-CSF treatment;
4. History of ≥ Grade 2 autoimmune reactions, allergic reactions or urticaria or other OncoVEX^GM-CSF-related non-hematological toxicities while on OncoVEX^GM-CSF treatment that required a dose delay or discontinuation of OncoVEX^GM-CSF therapy;
5. Symptomatic malignant disease progression that required alternative melanoma treatment;
6. Primary malignancy disease progression despite treatment with OncoVEX^GM-CSF;
7. Patient requested to be withdrawn from or was unable to comply with the demands of Study 002/03.
8. Patient was withdrawn from Study 002/03 at the discretion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, MD, Study Director — Amgen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Talimogene Laherparepvec
Started | 3
Completed | 2
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Talimogene Laherparepvec: Participants received talimogene laherparepvec 10⁸ PFU/mL (up to 4 mL depending on tumor size) administered intratumorally every 2 weeks, on Day 1 and Day 15 of 28-day cycles until discontinuation criteria were met.
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — Baseline measure data are from the beginning of the 002/03 study.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 2
    >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 62 [58 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 (Fully active) | 2
    1 (Restrictive but ambulatory) | 1
Tumor, Node, Metastasis (TNM) Disease Stage [Number; unit: participants] — Stage IIIC: Ulcerated lesion and 1 lymph node with macrometastasis; 2-3 nodes with macrometastasis or ≥ 4 metastatic lymph nodes, matted lymph nodes, or in-transit met(s)/satellite(s); Stage IV: M1a: Spread to skin, subcutaneous tissue, or lymph nodes; normal lactate dehydrogenase (LDH) level; M1b: Spread to lungs; normal LDH level; M1c: Spread to all other visceral organs, normal LDH level or any distant disease with elevated LDH level.
  participants
    Stage IIIC | 1
    Stage IVM1a | 1
    Stage IVM1b | 0
    Stage IVM1c | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The severity of an adverse event (AE) was graded according to Common Toxicity Criteria for Adverse Events (CTCAE) Version 3 (1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death).
  Serious adverse events include death, life-threatening events, events requiring or prolonging hospitalization, result in persistent or significant disability/incapacity, or a congenital anomaly/birth defect, or otherwise important medical events that may jeopardise the patient or require intervention to prevent one of the above outcomes.
Time Frame: From the first dose of talimogene laherparepvec in Study 002-03-E and within 30 days of the last dose; median duration of treatment was 267 days.
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 3
participants
  Any adverse event | 3
  Treatment-related adverse event | 3
  Adverse event ≥ grade 3 | 0
  Fatal adverse events | 0
  Serious adverse events | 0
  Discontinued study treatment due to adverse event | 0

2. Secondary Outcome: Number of Participants With an Objective Response
Description: Objective response is defined as participants with an overall best response of complete response or partial response. The objective response to treatment was assessed by computed tomography (CT) scanning or other clinical measurement using modified Response Evaluation Criteria In Solid Tumors (RECIST).
  Responses must have been confirmed two visits not less than 4 weeks apart.
  Tumor burden for a visit was calculated as the sum of the longest diameters of all tumors identified and measured up to that visit. Tumor response at each visit was derived from tumor burden, as follows:
  * Complete response (CR): zero tumor burden
  * Partial response (PR): a 30% or greater decrease in tumor burden
  * Progressive disease (PD): a 20% or greater increase in tumor burden
  * Stable disease (SD): none of the above (a < 30% decrease and < 20% increase in tumor burden)
Time Frame: Every 12 weeks from the start of therapy in this extension protocol, or 12 weeks from the last assessment in the 002/03 protocol (whichever date is later) through 30 days after administration of the last dose; median duration of treatment was 267 days.
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 3
participants | 2

3. Secondary Outcome: Number of Participants Alive at the Time of Study Discontinuation or Completion
Time Frame: At end of study, median duration of treatment was 267 days
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Time Frame: From the first dose of talimogene laherparepvec in Study 002-03-E and within 30 days of the last dose; median duration of treatment was 267 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Talimogene Laherparepvec
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=3)
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Lip swelling (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.